CLINICAL TRIAL: NCT00139984
Title: Impact of Ambulatory Blood Pressure Monitoring for Antihypertensive Treatment Guidance in Medical Outpatients: The Hyper-ABC Study
Brief Title: Ambulatory Blood Pressure Monitoring for Antihypertensive Treatment Guidance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EKBB183/03
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Hypertension; Ambulatory blood pressure monitoring; Blood pressure; Risk assessment
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: 24 hour blood pressure measurement

SUMMARY:
The purpose of this study is to determine whether in patients with arterial hypertension, treatment guidance using 24-hour blood pressure measurement results in better blood pressure control compared to treatment guidance using office blood pressure measurement.

DETAILED DESCRIPTION:
Blood pressure control in arterial hypertension remains poor, despite the availability of effective drug treatment. Therefore, strategies to increase blood pressure control are urgently needed. 24 hour blood pressure is a better predictor of cardiovascular morbidity and mortality than office blood pressure. Furthermore, the lower variability of measurements over time of 24 hour blood pressure could allow better adjustment of antihypertensive therapy. However, there are only scarce data about antihypertensive treatment adjustment using 24 hour blood pressure instead of office blood pressure.

Aim: To test the hypothesis that a 24 hour blood pressure guided therapy is is more effective in reaching blood pressure control when compared to conventional office blood pressure guided therapy.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled hypertension (office BP >139/89mmHg AND 24h BP >129/79mmHg)

Exclusion Criteria:

* Severe concomitant illness including heart failure, significant valvular heart disease or malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2003-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour systolic blood pressure from baseline to 1 year

SECONDARY OUTCOMES:
Change in 24-hour diastolic blood pressure from baseline to 1 year
Primary outcome measure in patients with treated hypertension at baseline

CONTACTS AND LOCATIONS:
Overall Officials: David Conen, MD, Principal Investigator — Cardiology, University Hospital Basel
Locations (2):
- Switzerland (2):
  - Medical Outpatient Clinic, University Hospital Basel, Basel
  - Private Practice, Basel

REFERENCES:
- [Derived] Conen D, Tschudi P, Martina B. Twenty-four hour ambulatory blood pressure for the management of antihypertensive treatment: a randomized controlled trial. J Hum Hypertens. 2009 Feb;23(2):122-9. doi: 10.1038/jhh.2008.106. Epub 2008 Aug 28. PMID 18754021